CLINICAL TRIAL: NCT04256629
Title: A Single-Centre, Randomised, Double-Blind, Placebo-Controlled, 3-Period, Cross-Over Phase I Study to Investigate the Effect on the QTcF Interval of a Single Dose of 2 Different Doses of Verinurad, Each in Combination With Allopurinol 300 mg, Compared With Placebo In Healthy Volunteers
Brief Title: A Study to Assess the Effect of Verinurad on the Electric Activity of the Heart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D5495C00012
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Results first posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers (Intended Indication: Chronic Kidney Disease)
Keywords: Randomised; Double-Blind; Placebo-Controlled; 3-Period Crossover; Verinurad; Allopurinol; Phase 1
MeSH Terms: interventions — verinurad; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is double-blind with regards to treatment (verinurad and allopurinol or the matching placebos) at each dose level. Placebo will be matched with verinurad and allopurinol for appearance and amount. Subjects randomized to placebo will receive the same volume of oral suspension as subjects on active drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment ABC (Experimental): Subjects will receive a single dose of all 3 treatments (A, B, and C) in a crossover design with wash-out periods of at least 7 days between each study dose administration.
  Interventions: Drug: Verinurad; Drug: Placebo; Drug: Allopurinol
- Treatment BCA (Experimental): Subjects will receive a single dose of all 3 treatments (B, C, and A) in a crossover design with wash-out periods of at least 7 days between each study dose administration.
  Interventions: Drug: Verinurad; Drug: Placebo; Drug: Allopurinol
- Treatment CAB (Experimental): Subjects will receive a single dose of all 3 treatments (C, A, and B) in a crossover design with wash-out periods of at least 7 days between each study dose administration.
  Interventions: Drug: Verinurad; Drug: Placebo; Drug: Allopurinol
- Treatment ACB (Experimental): Subjects will receive a single dose of all 3 treatments (A, C, and B) in a crossover design with wash-out periods of at least 7 days between each study dose administration.
  Interventions: Drug: Verinurad; Drug: Placebo; Drug: Allopurinol
- Treatment BAC (Experimental): Subjects will receive a single dose of all 3 treatments (B, A, and C) in a crossover design with wash-out periods of at least 7 days between each study dose administration.
  Interventions: Drug: Verinurad; Drug: Placebo; Drug: Allopurinol
- Treatment CBA (Experimental): Subjects will receive a single dose of all 3 treatments (C, B and A) in a crossover design with wash-out periods of at least 7 days between each study dose administration.
  Interventions: Drug: Verinurad; Drug: Placebo; Drug: Allopurinol

INTERVENTIONS:
Drug: Verinurad — Randomized subjects will receive oral dose of verinurad
  Other Names: verinurad ER 24 mg; verinurad IR 40 mg
Drug: Placebo — Randomized subjects will receive oral dose of placebo
  Other Names: verinurad matching placebo; allopurinol matching placebo
Drug: Allopurinol — Randomized subjects will receive oral dose of allpurinol (Treatment A and B)
  Other Names: allopurinol 300 mg

SUMMARY:
This study will be conducted to investigate the safety of verinurad in healthy volunteers in combination with allopurinol 300 mg, compared with placebo in particular its effect on electrocardiogram (ECG), with focus on the QT/QTc interval

DETAILED DESCRIPTION:
This study will be conducted as a single-centre, randomised, placebo-controlled, double-blind, 3-period, crossover study to assess the effect on the QTcF interval of a single oral dose of verinurad 24 mg extended release (ER8) formulation (therapeutic exposure) or verinurad 40 mg immediate release (IR) formulation (supra-therapeutic exposure), each in combination with allopurinol 300 mg, compared to placebo in healthy subjects.

There are 3 study treatments:

* Treatment A: Verinurad 24 mg ER8 formulation co-administered with 300 mg allopurinol
* Treatment B: Verinurad 40 mg IR formulation co-administered with 300 mg allopurinol
* Treatment C: Matched placebos for both verinurad and allopurinol

All subjects will receive a single dose of all 3 treatments (A, B, and C) in a cross-over design with wash-out periods of at least 7 days between each study dose administration.

Subjects will be randomised to the treatment sequence (ABC, BCA, CAB, etc.) using William's Latin square. The treatments will be administered in a double-blind manner after an overnight fast of at least 10 hours.

The study will comprise the following periods (visits):

* Screening Period of maximum 28 days (Visit 1);
* Three treatment periods of 3 days each, during which subjects will be resident at the study centre from the morning of the day before administration of the study dose until discharge 2 days after study dose administration (Visits 2 to 4);
* Wash-out periods of at least 7 days between each study dose administration;
* Final visit within 7 to 10 days after the last study dose administration (Visit 5).

Each subject will be involved in the study for approximately 53 days and have 5 study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study-specific procedures.
2. Healthy male and female subjects aged 18 to 50 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at Screening and on admission to the study centre must be:

(1) Not pregnant or currently lactating or breast-feeding. (2) Of non-childbearing potential confirmed at the Screening Visit by fulfilling one of the following criteria: (i) Post-menopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the post-menopausal range (FSH >40 IU/mL).

(ii) Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

(3) OR, if of childbearing potential, must be willing to use an acceptable method of contraception to avoid pregnancy for the entire study period and 3 months after the Follow-up Visit.

4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

5. Serum uric acid (sUA) <300 μmol/L at Screening (Visit 1) and sUA <330 μmol/L on Day -1 in every treatment period (Visit 2 to 4). Note: Since sUA levels might vary on a daily basis, subjects with sUA ≥330 μmol/L on Day -1 will be retested. Treatment on Day 1 will only be administered when the sUA level on Day -1 is <330 μmol/L upon retesting. Subjects with sUA ≥330 μmol/L despite retesting, may conduct the treatment period at a later date when they have sUA <330 μmol/L.

6. Must be able to swallow multiple capsules/tablets.

Exclusion criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
4. Subject has a positive test result for SARS-CoV-2 RT-PCR before randomisation.
5. Subject has clinical signs and symptoms consistent with COVID-19, eg, fever, dry cough, dyspnoea, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
6. History of severe COVID-19 (hospitalization, extracorporeal membrane oxygenation, mechanically ventilated).
7. Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, at Screening (Visit 1) as judged by the Investigator, including:

(1) Alanine aminotransferase (ALT) >1.5 × upper limit of normal (ULN) (2) Aspartate aminotransferase (AST) >1.5 × ULN (3) Bilirubin (total) >1.5 × ULN (4) Gamma glutamyl transpeptidase (GGT) >1.5 × ULN 8. Any clinically significant abnormal findings in vital signs at Screening as judged by the Investigator, including:

(1) Systolic blood pressure <90 mmHg or >140 mmHg (2) Diastolic blood pressure <50 mmHg or >90 mmHg (3) Heart rate <50 or >90 bpm 9. Carrier of the HLA-B*58:01 allele. 10. Any clinically important abnormalities in rhythm, conduction or morphology of the 12 lead safety ECG and any clinically important abnormalities in the 12-lead safety ECG as considered by the Investigator that may interfere with the interpretation of QT interval corrected for heart rate using Fridericia's formula (QTcF), including abnormal ST T wave morphology, particularly in the Clinical Study Protocol (CSP)-defined primary lead for dECG analysis or left ventricular hypertrophy:

1. Prolonged QTcF >450 ms or shortened QTcF <340 ms or family history of long QT syndrome.
2. PR (PQ) interval shortening <120 ms (PR >110 ms but <120 ms is acceptable if there is no evidence of ventricular pre-excitation).
3. PR (PQ) interval prolongation (>220 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation.
4. Persistent or intermittent complete bundle branch block, incomplete bundle branch block, or intraventricular conduction delay with QRS >110 ms. Subjects with QRS >110 ms but <115 ms are acceptable if there is no evidence of ventricular hypertrophy or pre-excitation.

11. Any positive result on Screening for serum hepatitis B surface antigen OR anti-HBc antibody, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.

12. Suspected or known Gilbert's syndrome. 13. Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the 3 months prior to Screening.

14. Known or suspected history of alcohol abuse or excessive intake of alcohol as judged by the Investigator. Excessive intake of alcohol defined as the regular consumption of more than 24 g of alcohol per day for men or 12 g per day for women.

15. Positive screen for drugs of abuse, cotinine (nicotine) or alcohol at the Screening Visit or on each admission to the study centre.

16. Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) as judged by the Investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (eg, >5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the study site.

17. Previous hypersensitivity reaction to allopurinol or any URAT1 inhibitor. 18. Subjects who are pregnant, breast-feeding or planning to become pregnant (pregnancy is to be avoided for the entire study period and 3 months after the Follow up Visit).

19. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.

20. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 × the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or within 5 half-lives (whichever is longer). Hormone replacement therapy is allowed for females.

21. Plasma donation within 1 month of Screening or any blood donation/blood loss >500 mL during the 3 months prior to Screening.

22. Has received another new chemical or biological entity (defined as a compound which has not been approved for marketing in the US) within 30 days or within 5 half lives (whichever is longer) of the first administration of IMP in this study.

Note: Subjects consented and screened, but not randomised in this study or a previous Phase I study, are not excluded.

23. Involvement of any AstraZeneca, Parexel or study site employee or their close relatives.

24. Subjects who have previously received verinurad. 25. Subjects who cannot communicate reliably with the Investigator and/or are not able to read, speak and understand the German language.

26. Judgment by the Investigator that the subject should not participate in the study if there are any ongoing or recent (ie, during the Screening Period) minor medical complaints that may interfere with the interpretation of the study data or are considered unlikely to comply with study procedures, restrictions and requirements.

27. Subjects who are vegans or have medical dietary restrictions. 28. Vulnerable subjects, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

29. Subjects who are regularly exposed to COVID-19 (eg, health care professionals working in COVID-19 wards or at emergency departments) as part of their daily life.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kӧrnicke, MD, Principal Investigator — PAREXEL Early Phase Clinical Unit Berlin
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Parkinson J, Dota C, Kallgren C, Gottfridsson C, Bjursell M, Perl S, Kӧrnicke T, Rekic D, Johansson S. Verinurad does not prolong QTc interval: a thorough QT study using concentration-QTc modelling. Br J Clin Pharmacol. 2023 Jun;89(6):1747-1755. doi: 10.1111/bcp.15637. Epub 2023 Jan 2. PMID 36504291
- See also: Protocol and Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5495C00012&attachmentIdentifier=26cfccca-107f-485c-bed6-d233c134942d&fileName=D5495C00012_Protocol__Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5495C00012&attachmentIdentifier=776039fd-c263-47a0-a196-114fde71dd4f&fileName=D5495C00012_CSR_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 24 healthy male and female participants at a single study center - Parexel Early Phase Clinical Unit (Berlin).
Pre-assignment Details: The study consisted of a Screening Period of maximum 28 days. There were wash-out periods of at least 7 days between each study dose administration. The assessments were done as per the schedule of assessment.
Groups:
- Treatment Sequence ABC: Randomised participants received single doses of all 3 study treatments (Treatment A: Verinurad 24 mg extended release [ER8] formulation co-administered with 300 mg allopurinol, Treatment B: Verinurad 40 mg immediate release [IR] formulation co-administered with 300 mg allopurinol, and Treatment C: Matching placebos for both verinurad and allopurinol) in a cross-over design with wash-out periods of at least 7 days between each study dose administration under fasted conditions.
- Treatment Sequence BCA: Randomised participants received single doses of all 3 study treatments (Treatment B: Verinurad 40 mg IR formulation co-administered with 300 mg allopurinol, Treatment C: Matching placebos for both verinurad and allopurinol, and Treatment A: Verinurad 24 mg ER8 formulation co-administered with 300 mg allopurinol) in a cross-over design with wash-out periods of at least 7 days between each study dose administration under fasted conditions.
- Treatment Sequence CAB: Randomised participants received single doses of all 3 study treatments (Treatment C: Matching placebos for both verinurad and allopurinol, Treatment A: Verinurad 24 mg ER8 formulation co-administered with 300 mg allopurinol, and Treatment B: Verinurad 40 mg IR formulation co-administered with 300 mg allopurinol) in a cross-over design with wash-out periods of at least 7 days between each study dose administration under fasted conditions.
- Treatment Sequence ACB: Randomised participants received single doses of all 3 study treatments ( Treatment A: Verinurad 24 mg ER8 formulation co-administered with 300 mg allopurinol, Treatment C: Matching placebos for both verinurad and allopurinol, and Treatment B: Verinurad 40 mg IR formulation co-administered with 300 mg allopurinol) in a cross-over design with wash-out periods of at least 7 days between each study dose administration under fasted conditions.
- Treatment Sequence BAC: Randomised participants received single doses of all 3 study treatments (Treatment B: Verinurad 40 mg IR formulation co-administered with 300 mg allopurinol, Treatment A: Verinurad 24 mg ER8 formulation co-administered with 300 mg allopurinol, and Treatment C: Matching placebos for both verinurad and allopurinol) in a cross-over design with wash-out periods of at least 7 days between each study dose administration under fasted conditions.
- Treatment Sequence CBA: Randomised participants received single doses of all 3 study treatments (Treatment C: Matching placebos for both verinurad and allopurinol, Treatment B: Verinurad 40 mg IR formulation co-administered with 300 mg allopurinol, and Treatment A: Verinurad 24 mg ER8 formulation co-administered with 300 mg allopurinol) in a cross-over design with wash-out periods of at least 7 days between each study dose administration under fasted conditions.
Period: Overall Study
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence CBA
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 3 | 4 | 4 | 4 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence CBA | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (13.35) | 30.0 (6.16) | 32.8 (14.08) | 35.5 (7.14) | 31.0 (12.25) | 34.0 (12.36) | 33.7 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 1 | 0 | 5
  Male | 3 | 3 | 3 | 3 | 3 | 4 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 4 | 4 | 3 | 4 | 3 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Model Predicted Baseline-corrected and Placebo-corrected QT Interval Corrected for Heart Rate (HR) Using Fridericia's Formula (QTcF)(ΔΔQTcF) (Derived From Concentration-QTcF Analysis) at Geometric Mean of Cmax of Verinurad
Description: Assessment of the effect of a single dose of verinurad given as either a 24 mg ER8 formulation (clinical exposure) or a 40 mg IR formulation (exposure needed to waive positive control as per question 5.1 of International Council for Harmonisation Guideline E14 and associated Questions and Answers [ICH E14 Q&A]), both in combination with allopurinol 300 mg, on the QTcF interval compared to placebo using a concentration-QTcF analysis.
  A linear mixed-effect concentration-QTcF model was used as the primary analysis. This is a result of the statistical model so it does not have values for every timepoint, it is just one set of numbers - summarizes data across all timepoints. No non-placebo-corrected QTcF data values were collected or could be obtained for each Arm/Group at Cmax of Verinurad.
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: In the Primary Outcome we present the predicted value of ΔΔQTcF based on a statistical model created for the study. The results may be presented for the active arms only, since the placebo arm did not receive Verinurad and thus have no Cmax. Placebo-corrected and baseline adjusted QTcF, ∆∆QTcF with 90% confidence interval at the verinurad maximum concentration of interest is presented as the primary result from the analysis.
Measure: Geometric Mean (90% Confidence Interval); unit: msec
Groups:
- Treatment A: Participants received a single dose of verinurad 24 mg ER8 formulation co-administered with 300 mg allopurinol
- Treatment B: Participants received a single dose of verinurad 40 mg IR formulation co-administered with 300 mg allopurinol
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 24 | 24
msec | -2.8 [-4.7 to -0.9] | -0.3 [-3.1 to 2.5]

2. Secondary Outcome: Baseline-corrected Heart Rate (ΔHR)
Description: Investigation of the effect of verinurad given either as a 24 mg ER8 formulation (clinical exposure) or a 40 mg IR formulation (exposure needed to waive positive control as per question 5.1 of ICH E14 Q&A), both in combination with allopurinol 300 mg, on heart rate (HR).
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hour (h) post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: The PD Analysis Set consisted of all participants in the Safety Analysis Set for whom baseline and post-baseline QTcF results from smoothed dECG data were available for at least 1 treatment period and who had no major protocol deviations thought to impact the analysis of the dECG data. Here, number analyzed in each row signifies only the participants with available data that were analyzed for that particular day and time.
Measure: Mean (95% Confidence Interval); unit: Beats per minute (bpm)
Groups:
- Treatment C: Participants received matching placebos for both verinurad and allopurinol
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
Beats per minute (bpm)
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 0.5 h | -0.8 [-1.7 to 0.1] | -2.0 [-3.2 to -0.7] | -0.5 [-1.8 to 0.8]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1 h | -0.9 [-2.0 to 0.3] | -1.0 [-2.2 to 0.1] | 0.1 [-1.4 to 1.6]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1.5 h | -2.3 [-3.8 to -0.7] | -1.3 [-2.5 to -0.2] | -0.6 [-1.9 to 0.8]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 2 h | -1.9 [-3.5 to -0.3] | -2.5 [-4.0 to -1.0] | -0.5 [-1.9 to 1.0]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 3 h | -0.8 [-2.8 to 1.2] | -1.7 [-3.3 to -0.1] | 0.6 [-0.9 to 2.1]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 4 h | 9.3 [6.2 to 12.4] | 7.2 [4.9 to 9.4] | 8.7 [6.2 to 11.2]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 5 h | 6.4 [3.9 to 8.8] | 5.8 [3.0 to 8.5] | 6.2 [4.0 to 8.4]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 6 h | 2.8 [0.6 to 4.9] | 2.3 [0.3 to 4.4] | 4.1 [2.4 to 5.7]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 8 h | 9.6 [8.0 to 11.3] | 6.5 [4.6 to 8.3] | 8.5 [6.4 to 10.6]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 12 h | 0.3 [-1.4 to 1.9] | 0.8 [-0.7 to 2.4] | 2.3 [0.2 to 4.4]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 24 h | 0.0 [-1.9 to 1.9] | 1.4 [-0.2 to 3.0] | 0.9 [-1.0 to 2.8]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 36 h | 9.1 [5.5 to 12.8] | 9.6 [7.0 to 12.3] | 9.5 [6.0 to 13.0]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 24 | 23
  Day 3/ 48 h | 4.9 [2.0 to 7.8] | 3.9 [2.0 to 5.8] | 5.3 [3.2 to 7.3]

3. Secondary Outcome: Baseline-corrected and Placebo-adjusted Heart Rate (ΔΔHR)
Description: Investigation of the effect of verinurad given either as a 24 mg ER8 formulation (clinical exposure) or a 40 mg IR formulation (exposure needed to waive positive control as per question 5.1 of ICH E14 Q&A), both in combination with allopurinol 300 mg, on HR.
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: bpm
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 24 | 24
bpm
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 0.5 h | -0.4 [-2.0 to 1.2] | -1.4 [-3.2 to 0.4]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1 h | -0.9 [-2.8 to 1.0] | -1.1 [-3.0 to 0.7]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1.5 h | -1.6 [-3.5 to 0.3] | -0.7 [-2.7 to 1.3]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 23
  Day 1/ 2 h | -1.3 [-3.1 to 0.6] | -1.8 [-3.9 to 0.2]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 23
  Day 1/ 3 h | -1.5 [-3.1 to 0.1] | -2.2 [-4.2 to -0.2]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 23
  Day 1/ 4 h | 0.5 [-1.7 to 2.6] | -1.4 [-3.6 to 0.8]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 5 h | 0.1 [-2.7 to 3.0] | -0.3 [-3.7 to 3.0]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 23
  Day 1/ 6 h | -1.2 [-3.4 to 0.9] | -1.6 [-3.9 to 0.7]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 23
  Day 1/ 8 h | 1.0 [-1.3 to 3.3] | -2.0 [-5.0 to 1.1]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 23
  Day 1/ 12 h | -2.1 [-4.6 to 0.4] | -1.4 [-4.1 to 1.3]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 23
  Day 2/ 24 h | -0.9 [-2.2 to 0.5] | 0.7 [-1.6 to 3.0]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 23
  Day 2/ 36 h | -0.5 [-3.0 to 2.0] | 0.5 [-2.4 to 3.4]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 23
  Day 3/ 48 h | -0.4 [-2.6 to 1.9] | -1.1 [-3.8 to 1.5]

4. Secondary Outcome: Baseline-corrected RR Interval (ΔRR Interval)
Description: Investigation of the effect of verinurad given either as a 24 mg ER8 formulation (clinical exposure) or a 40 mg IR formulation (exposure needed to waive positive control as per question 5.1 of ICH E14 Q&A), both in combination with allopurinol 300 mg, on additional dECG variable (RR).
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Milli second (msec)
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
Milli second (msec)
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 0.5 h | 13.6 [-2.1 to 29.3] | 28.2 [9.2 to 47.2] | 6.7 [-17.3 to 30.7]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1 h | 14.8 [-8.8 to 38.5] | 15.8 [-4.8 to 36.3] | -8.3 [-35.6 to 19.1]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1.5 h | 47.1 [15.1 to 79.2] | 20.3 [5.3 to 35.3] | 6.4 [-17.7 to 30.4]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 2 h | 35.6 [7.7 to 63.6] | 36.5 [14.5 to 58.4] | 6.9 [-15.6 to 29.4]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 3 h | 11.3 [-24.8 to 47.5] | 24.4 [0.2 to 48.7] | -12.2 [-37.7 to 13.2]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 4 h | -139.7 [-194.9 to -84.5] | -111.7 [-151.7 to -71.7] | -133.8 [-181.1 to -86.5]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 5 h | -98.8 [-145.5 to -52.1] | -82.6 [-122.6 to -42.6] | -101.9 [-143.3 to -60.5]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 6 h | -45.4 [-83.0 to -7.8] | -44.6 [-76.8 to -12.3] | -66.7 [-96.7 to -36.7]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 8 h | -143.9 [-173.4 to -114.4] | -100.6 [-129.8 to -71.4] | -128.7 [-165.1 to -92.4]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 12 h | -5.0 [-39.8 to 29.7] | -16.3 [-43.1 to 10.5] | -39.9 [-68.8 to -10.9]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 24 h | -1.8 [-35.1 to 31.5] | -20.9 [-45.3 to 3.5] | -17.4 [-50.6 to 15.7]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 36 h | -129.2 [-170.7 to -87.7] | -134.1 [-170.1 to -98.0] | -132.0 [-177.0 to -87.1]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 24 | 23
  Day 3/ 48 h | -76.0 [-118.5 to -33.4] | -63.2 [-91.2 to -35.1] | -81.3 [-113.3 to -49.4]

5. Secondary Outcome: Baseline-corrected and Placebo-adjusted RR Interval (ΔΔRR Interval)
Description: as for outcome 4
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 24 | 24
msec
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 0.5 h | 6.7 [-23.2 to 36.6] | 20.7 [-10.5 to 51.9]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1 h | 22.2 [-13.3 to 57.7] | 23.3 [-9.5 to 56.0]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1.5 h | 38.9 [-1.2 to 79.0] | 13.0 [-15.3 to 41.2]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 23
  Day 1/ 2 h | 26.9 [-6.3 to 60.0] | 26.9 [-2.2 to 55.9]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 23
  Day 1/ 3 h | 25.1 [-7.2 to 57.4] | 35.1 [5.7 to 64.4]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 23
  Day 1/ 4 h | -3.4 [-36.4 to 29.6] | 18.8 [-12.8 to 50.4]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 5 h | 4.6 [-44.5 to 53.8] | 17.8 [-33.8 to 69.5]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 23
  Day 1/ 6 h | 21.0 [-16.1 to 58.2] | 19.7 [-8.7 to 48.2]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 23
  Day 1/ 8 h | -12.8 [-46.7 to 21.1] | 25.9 [-14.5 to 66.3]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 23
  Day 1/ 12 h | 36.5 [-4.9 to 78.0] | 22.1 [-18.6 to 62.9]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 23
  Day 2/ 24 h | 15.1 [-13.9 to 44.2] | -6.8 [-42.1 to 28.6]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 23
  Day 2/ 36 h | 5.7 [-26.0 to 37.3] | -7.1 [-50.7 to 36.6]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 23
  Day 3/ 48 h | 6.5 [-29.9 to 42.9] | 14.8 [-23.9 to 53.4]

6. Secondary Outcome: Baseline-corrected PR Interval (ΔPR Interval)
Description: Investigation of the effect of verinurad given either as a 24 mg ER8 formulation (clinical exposure) or a 40 mg IR formulation (exposure needed to waive positive control as per question 5.1 of ICH E14 Q&A), both in combination with allopurinol 300 mg, on additional dECG variable (PR).
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
msec
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 0.5 h | -1.3 [-2.8 to 0.2] | -0.9 [-2.7 to 1.0] | -0.8 [-2.0 to 0.3]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1 h | -0.4 [-2.3 to 1.5] | -1.3 [-3.1 to 0.5] | -0.7 [-1.6 to 0.3]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1.5 h | -1.8 [-4.1 to 0.5] | -0.6 [-2.5 to 1.3] | -0.8 [-2.2 to 0.5]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 2 h | -1.2 [-3.6 to 1.1] | -1.7 [-4.2 to 0.7] | 0.2 [-1.2 to 1.6]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 3 h | 0.1 [-1.7 to 1.9] | -1.3 [-3.2 to 0.7] | -1.6 [-3.1 to -0.1]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 4 h | -3.5 [-6.4 to -0.5] | -3.2 [-5.7 to -0.7] | -2.7 [-6.1 to 0.6]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 5 h | -4.0 [-6.3 to -1.6] | -4.5 [-7.0 to -2.0] | -3.6 [-6.6 to -0.6]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 6 h | -4.6 [-6.1 to -3.1] | -2.2 [-4.9 to 0.5] | -2.6 [-4.7 to -0.4]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 8 h | -6.1 [-9.4 to -2.8] | -5.8 [-8.4 to -3.1] | -5.6 [-8.8 to -2.3]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 12 h | -1.0 [-3.9 to 1.8] | -0.9 [-3.3 to 1.5] | -1.0 [-4.1 to 2.2]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 24 h | -1.0 [-3.6 to 1.5] | -0.5 [-2.5 to 1.5] | -1.0 [-3.4 to 1.3]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 36 h | 0.5 [-2.6 to 3.5] | 0.8 [-2.2 to 3.7] | -2.4 [-6.5 to 1.7]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 24 | 23
  Day 3/ 48 h | -0.7 [-3.4 to 1.9] | 0.4 [-2.7 to 3.6] | -0.7 [-3.3 to 1.8]

7. Secondary Outcome: Baseline-corrected and Placebo-adjusted PR Interval (ΔΔPR Interval)
Description: as for outcome 6
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 24 | 24
msec
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 0.5 h | -0.5 [-2.2 to 1.3] | 0.0 [-2.1 to 2.1]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1 h | 0.3 [-1.6 to 2.2] | -0.3 [-1.9 to 1.2]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1.5 h | -0.7 [-3.2 to 1.8] | 0.5 [-1.7 to 2.7]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 23
  Day 1/ 2 h | -1.3 [-3.8 to 1.3] | -1.7 [-4.1 to 0.7]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 23
  Day 1/ 3 h | 1.7 [-0.6 to 4.1] | 0.4 [-2.4 to 3.2]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 23
  Day 1/ 4 h | -0.3 [-3.1 to 2.5] | 0.2 [-2.6 to 2.9]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 5 h | 0.1 [-3.2 to 3.4] | -0.3 [-3.0 to 2.4]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 23
  Day 1/ 6 h | -1.7 [-3.7 to 0.3] | 0.4 [-2.4 to 3.2]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 23
  Day 1/ 8 h | -0.1 [-3.3 to 3.1] | 0.2 [-2.7 to 3.1]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 23
  Day 1/ 12 h | -0.0 [-2.7 to 2.6] | 0.3 [-2.5 to 3.1]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 23
  Day 2/ 24 h | -0.0 [-2.9 to 2.8] | 0.5 [-2.0 to 3.0]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 23
  Day 2/ 36 h | 3.1 [-1.3 to 7.5] | 2.8 [-1.7 to 7.3]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 23
  Day 3/ 48 h | 0.2 [-2.8 to 3.2] | 0.9 [-1.7 to 3.5]

8. Secondary Outcome: Baseline-corrected QRS Interval (ΔQRS Interval)
Description: Investigation of the effect of verinurad given either as a 24 mg ER8 formulation (clinical exposure) or a 40 mg IR formulation (exposure needed to waive positive control as per question 5.1 of ICH E14 Q&A), both in combination with allopurinol 300 mg, on additional dECG variable (QRS).
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
msec
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 0.5 h | -0.5 [-1.2 to 0.3] | -0.6 [-1.6 to 0.4] | 0.0 [-0.6 to 0.6]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1 h | -0.7 [-1.4 to -0.0] | -0.9 [-1.8 to -0.0] | 0.1 [-0.5 to 0.8]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1.5 h | -0.5 [-1.4 to 0.5] | -0.5 [-1.2 to 0.2] | 0.3 [-0.3 to 1.0]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 2 h | 0.0 [-1.1 to 1.1] | -0.8 [-1.8 to 0.2] | 0.3 [-0.4 to 1.1]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 3 h | -0.6 [-1.7 to 0.4] | -0.8 [-1.9 to 0.2] | -0.4 [-1.2 to 0.3]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 4 h | 1.3 [0.6 to 2.1] | 1.2 [-0.3 to 2.7] | 1.7 [0.8 to 2.7]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 5 h | -0.3 [-1.3 to 0.6] | -0.6 [-1.9 to 0.7] | 0.1 [-1.2 to 1.3]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 6 h | -1.2 [-1.9 to -0.5] | -1.3 [-2.2 to -0.3] | -0.7 [-1.9 to 0.5]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 8 h | -2.6 [-3.7 to -1.6] | -2.5 [-3.4 to -1.6] | -1.7 [-3.3 to 0.0]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 12 h | -0.5 [-1.2 to 0.3] | -0.9 [-2.0 to 0.2] | -0.4 [-1.4 to 0.7]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 24 h | -1.1 [-1.8 to -0.3] | -1.3 [-2.0 to -0.5] | -0.9 [-1.8 to -0.0]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 36 h | -0.6 [-1.4 to 0.2] | -0.8 [-2.0 to 0.4] | -0.7 [-1.9 to 0.4]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 24 | 23
  Day 3/ 48 h | -1.0 [-1.8 to -0.1] | -0.7 [-1.4 to 0.1] | -0.7 [-1.6 to 0.2]

9. Secondary Outcome: Baseline-corrected and Placebo-corrected QRS Interval (ΔΔQRS Interval)
Description: as for outcome 8
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 24 | 24
msec
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 0.5 h | -0.4 [-1.2 to 0.4] | -0.7 [-1.7 to 0.4]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1 h | -0.9 [-1.7 to 0.0] | -1.1 [-2.1 to -0.1]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1.5 h | -0.8 [-1.8 to 0.1] | -0.8 [-1.8 to 0.1]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 23
  Day 1/ 2 h | -0.4 [-1.5 to 0.8] | -1.2 [-2.2 to -0.1]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 23
  Day 1/ 3 h | -0.2 [-1.3 to 0.9] | -0.4 [-1.8 to 1.0]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 23
  Day 1/ 4 h | -0.4 [-1.4 to 0.6] | -0.7 [-2.3 to 0.8]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 5 h | -0.4 [-1.9 to 1.1] | -0.8 [-2.4 to 0.7]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 23
  Day 1/ 6 h | -0.5 [-1.7 to 0.7] | -0.6 [-2.0 to 0.9]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 23
  Day 1/ 8 h | -1.0 [-2.5 to 0.6] | -0.9 [-2.7 to 0.9]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 23
  Day 1/ 12 h | 0.0 [-1.2 to 1.2] | -0.6 [-2.0 to 0.9]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 23
  Day 2/ 24 h | -0.1 [-1.1 to 1.0] | -0.3 [-1.5 to 0.9]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 23
  Day 2/ 36 h | 0.1 [-1.2 to 1.5] | -0.0 [-1.8 to 1.7]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 23
  Day 3/ 48 h | -0.2 [-1.4 to 1.0] | 0.0 [-1.2 to 1.3]

10. Secondary Outcome: Baseline-corrected QT Interval (ΔQT Interval)
Description: Investigation of the effect of verinurad given either as a 24 mg ER8 formulation (clinical exposure) or a 40 mg IR formulation (exposure needed to waive positive control as per question 5.1 of ICH E14 Q&A), both in combination with allopurinol 300 mg, on additional dECG variable (QT).
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
msec
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 0.5 h | 0.2 [-3.5 to 3.9] | 3.8 [0.3 to 7.4] | 0.4 [-2.8 to 3.6]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1 h | 1.5 [-1.7 to 4.7] | 4.5 [1.4 to 7.5] | 2.1 [-1.5 to 5.8]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1.5 h | 4.8 [-0.5 to 10.1] | 5.4 [1.8 to 9.0] | 3.7 [0.6 to 6.7]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 2 h | 5.0 [0.3 to 9.8] | 7.3 [4.3 to 10.3] | 5.3 [1.5 to 9.2]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 3 h | 2.1 [-2.2 to 6.5] | 4.5 [0.5 to 8.5] | 1.8 [-2.3 to 6.0]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 4 h | -19.9 [-27.2 to -12.6] | -12.7 [-19.0 to -6.4] | -15.6 [-20.9 to -10.4]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 5 h | -19.5 [-26.4 to -12.6] | -14.1 [-19.4 to -8.8] | -15.9 [-20.5 to -11.4]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 6 h | -16.0 [-21.9 to -10.2] | -11.0 [-15.8 to -6.1] | -12.7 [-17.2 to -8.2]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 8 h | -31.1 [-38.0 to -24.2] | -22.9 [-28.3 to -17.5] | -23.9 [-28.8 to -19.0]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 12 h | -0.7 [-6.0 to 4.5] | 0.3 [-5.2 to 5.8] | 0.3 [-4.9 to 5.4]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 24 h | -4.9 [-10.3 to 0.5] | -2.7 [-6.9 to 1.6] | -2.5 [-7.0 to 2.1]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 36 h | -24.8 [-33.6 to -16.0] | -24.1 [-29.1 to -19.1] | -21.6 [-29.4 to -13.8]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 24 | 23
  Day 3/ 48 h | -16.0 [-22.8 to -9.3] | -10.0 [-14.4 to -5.7] | -10.7 [-15.3 to -6.0]

11. Secondary Outcome: Baseline-corrected and Placebo-corrected QT Interval (ΔΔQT Interval)
Description: as for outcome 10
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 24 | 24
msec
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 0.5 h | -0.3 [-4.6 to 4.1] | 3.0 [-2.0 to 8.1]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1 h | -0.7 [-5.8 to 4.3] | 2.1 [-3.1 to 7.3]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1.5 h | 1.0 [-4.7 to 6.7] | 1.7 [-3.7 to 7.1]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 23
  Day 1/ 2 h | -0.7 [-5.8 to 4.4] | 1.7 [-3.5 to 6.8]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 23
  Day 1/ 3 h | 0.3 [-4.7 to 5.3] | 2.3 [-3.2 to 7.9]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 23
  Day 1/ 4 h | -4.3 [-8.7 to 0.0] | 2.1 [-3.2 to 7.4]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 5 h | -3.4 [-10.5 to 3.8] | 1.4 [-5.6 to 8.4]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 23
  Day 1/ 6 h | -3.6 [-9.1 to 1.9] | 1.7 [-3.1 to 6.6]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 23
  Day 1/ 8 h | -7.2 [-13.1 to -1.4] | 0.8 [-6.4 to 8.0]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 23
  Day 1/ 12 h | -0.8 [-7.1 to 5.5] | -0.4 [-8.0 to 7.2]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 23
  Day 2/ 24 h | -2.5 [-6.5 to 1.4] | -0.5 [-6.5 to 5.6]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 23
  Day 2/ 36 h | -3.3 [-8.4 to 1.8] | -3.0 [-10.2 to 4.3]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 23
  Day 3/ 48 h | -5.7 [-11.3 to -0.0] | 0.3 [-6.1 to 6.7]

12. Secondary Outcome: Baseline-corrected QTcF Interval (ΔQTcF Interval)
Description: Investigation of the effect of verinurad given either as a 24 mg ER8 formulation (clinical exposure) or a 40 mg IR formulation (exposure needed to waive positive control as per question 5.1 of ICH E14 Q&A), both in combination with allopurinol 300 mg, on additional dECG variable (QTcF).
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 24
msec
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 0.5 h | -1.7 [-4.6 to 1.3] | -0.3 [-2.3 to 1.7] | -0.5 [-2.3 to 1.2]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1 h | -0.4 [-1.7 to 0.9] | 2.3 [0.6 to 4.0] | 3.1 [1.2 to 5.0]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 1.5 h | -1.0 [-3.8 to 1.9] | 2.7 [-0.3 to 5.6] | 2.9 [1.2 to 4.6]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 2 h | 0.5 [-1.7 to 2.8] | 2.5 [0.7 to 4.3] | 4.6 [2.1 to 7.1]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 3 h | 0.7 [-2.1 to 3.5] | 1.2 [-0.9 to 3.3] | 3.3 [0.9 to 5.6]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 4 h | -0.6 [-4.2 to 2.9] | 2.3 [-2.4 to 7.0] | 2.7 [0.2 to 5.2]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 5 h | -6.3 [-9.1 to -3.6] | -2.5 [-6.6 to 1.6] | -2.5 [-5.2 to 0.3]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 6 h | -10.0 [-13.5 to -6.6] | -5.7 [-9.7 to -1.6] | -4.0 [-7.1 to -1.0]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 8 h | -12.1 [-16.7 to -7.5] | -10.0 [-14.2 to -5.9] | -7.0 [-10.6 to -3.4]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 24 | 23
  Day 1/ 12 h | 0.2 [-3.2 to 3.6] | 2.2 [-2.1 to 6.4] | 5.3 [2.1 to 8.5]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 24 h | -4.8 [-8.3 to -1.3] | 0.2 [-2.6 to 2.9] | 0.0 [-2.1 to 2.2]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 24 | 23
  Day 2/ 36 h | -7.6 [-12.6 to -2.6] | -6.1 [-10.0 to -2.1] | -3.7 [-7.5 to 0.2]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 24 | 23
  Day 3/ 48 h | -5.8 [-9.1 to -2.5] | -2.0 [-5.1 to 1.1] | 0.3 [-2.3 to 2.8]

13. Secondary Outcome: Baseline-corrected and Placebo-corrected QTcF Interval (ΔΔQTcF Interval)
Description: as for outcome 12
Time Frame: Baseline; Day 1: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 h post-dose; Day 2: 24 and 36 h post-dose; Day 3: 48 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 24 | 24
msec
  Day 1/ 0.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 0.5 h | -1.2 [-4.8 to 2.4] | -0.0 [-2.8 to 2.7]
  Day 1/ 1 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1 h | -3.4 [-5.7 to -1.0] | -0.9 [-3.5 to 1.8]
  Day 1/ 1.5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 1.5 h | -3.7 [-6.9 to -0.4] | -0.1 [-3.6 to 3.5]
  Day 1/ 2 h: number analyzed (Participants) | 22 | 23
  Day 1/ 2 h | -4.1 [-7.1 to -1.2] | -2.1 [-5.2 to 1.1]
  Day 1/ 3 h: number analyzed (Participants) | 22 | 23
  Day 1/ 3 h | -2.8 [-6.9 to 1.3] | -2.2 [-5.4 to 1.0]
  Day 1/ 4 h: number analyzed (Participants) | 22 | 23
  Day 1/ 4 h | -3.6 [-6.2 to -1.0] | -0.9 [-4.7 to 2.9]
  Day 1/ 5 h: number analyzed (Participants) | 22 | 23
  Day 1/ 5 h | -3.7 [-7.2 to -0.2] | -0.3 [-4.6 to 3.9]
  Day 1/ 6 h: number analyzed (Participants) | 22 | 23
  Day 1/ 6 h | -6.1 [-9.1 to -3.2] | -1.3 [-4.5 to 1.8]
  Day 1/ 8 h: number analyzed (Participants) | 22 | 23
  Day 1/ 8 h | -5.4 [-8.5 to -2.3] | -3.0 [-6.5 to 0.5]
  Day 1/ 12 h: number analyzed (Participants) | 22 | 23
  Day 1/ 12 h | -5.2 [-8.6 to -1.8] | -3.4 [-8.1 to 1.2]
  Day 2/ 24 h: number analyzed (Participants) | 22 | 23
  Day 2/ 24 h | -4.8 [-8.3 to -1.3] | 0.3 [-2.4 to 3.0]
  Day 2/ 36 h: number analyzed (Participants) | 22 | 23
  Day 2/ 36 h | -4.4 [-8.1 to -0.6] | -2.2 [-6.7 to 2.2]
  Day 3/ 48 h: number analyzed (Participants) | 22 | 23
  Day 3/ 48 h | -6.4 [-9.7 to -3.1] | -2.1 [-5.5 to 1.3]

14. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC) for Verinurad, M1, M8, Allopurinol, and Oxypurinol
Description: Assessment of the pharmacokinetic (PK) of verinurad and its metabolites (M1 and M8) and allopurinol and its metabolite (oxypurinol) in healthy participants.
Time Frame: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours post-dose; Day 2: 24 and 36 hours post-dose; Day 3: 48 hours post-dose
Population: The PK Analysis Set consisted of all participants in the Safety Analysis Set for whom at least 1 reportable PK parameter could be calculated and who had no major protocol deviations thought to impact the analysis of the PK data. Here, number analyzed in each row signifies only the participants with available data that were analyzed for Verinurad/M1/M8/allopurinol/oxypurinol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 22 | 24
h*ng/mL
  Verinurad: number analyzed (Participants) | 20 | 24
  Verinurad | 393.8 (34.99) | 918.7 (26.53)
  M1: number analyzed (Participants) | 21 | 24
  M1 | 413.7 (41.20) | 904.8 (34.49)
  M8: number analyzed (Participants) | 21 | 24
  M8 | 447.2 (32.30) | 895.0 (23.75)
  Allopurinol | 4501 (37.83) | 4617 (32.39)
  Oxypurinol | 151100 (16.74) | 145000 (17.02)

15. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC[0-t]) for Verinurad, M1, M8, Allopurinol, and Oxypurinol
Description: Assessment of the PK of verinurad and its metabolites (M1 and M8) and allopurinol and its metabolite (oxypurinol) in healthy participants.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 22 | 24
h*ng/mL
  Verinurad | 360.2 (32.95) | 880.4 (26.67)
  M1 | 383.2 (40.00) | 865.4 (35.23)
  M8 | 394.5 (30.32) | 847.8 (25.35)
  Allopurinol | 4408 (38.00) | 4524 (32.53)
  Oxypurinol | 136000 (15.67) | 131400 (15.12)

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Verinurad, M1, M8, Allopurinol, and Oxypurinol
Description: as for outcome 15
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 22 | 24
ng/mL
  Verinurad | 56.57 (36.34) | 459.7 (47.74)
  M1 | 54.92 (39.54) | 364.4 (48.92)
  M8 | 54.80 (31.28) | 297.8 (39.44)
  Allopurinol | 1610 (41.61) | 1780 (38.53)
  Oxypurinol | 7591 (16.77) | 7528 (20.28)

17. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) for Verinurad, M1, M8, Allopurinol, and Oxypurinol
Description: as for outcome 15
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 22 | 24
Hour
  Verinurad | 5.00 [3.00 to 12.00] | 1.02 [0.50 to 2.00]
  M1 | 5.00 [3.00 to 12.00] | 1.50 [1.00 to 2.00]
  M8 | 5.00 [4.00 to 12.00] | 1.50 [1.00 to 2.00]
  Allopurinol | 1.50 [0.50 to 3.00] | 1.50 [0.50 to 2.00]
  Oxypurinol | 5.00 [1.50 to 6.00] | 3.00 [1.50 to 5.00]

18. Secondary Outcome: Time Delay Between Drug Administration and the First Observed Concentration in Plasma (Tlag) for Verinurad, M1, M8, Allopurinol, and Oxypurinol
Description: as for outcome 15
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 22 | 24
Hour
  Verinurad | 0.50 [0.00 to 0.50] | 0.00 [0.00 to 0.00]
  M1 | 0.50 [0.00 to 1.00] | 0.00 [0.00 to 0.00]
  M8 | 0.50 [0.00 to 1.00] | 0.00 [0.00 to 0.00]
  Allopurinol | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 0.00]
  Oxypurinol | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

19. Secondary Outcome: Terminal Half-life (t½λz) for Verinurad, M1, M8, Allopurinol, and Oxypurinol
Description: as for outcome 15
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 22 | 24
Hour
  Verinurad: number analyzed (Participants) | 20 | 24
  Verinurad | 14.92 (5.355) | 13.33 (5.705)
  M1: number analyzed (Participants) | 21 | 24
  M1 | 14.30 (4.991) | 12.65 (4.354)
  M8: number analyzed (Participants) | 21 | 24
  M8 | 16.89 (8.832) | 13.96 (4.065)
  Allopurinol | 1.020 (0.2327) | 1.012 (0.1090)
  Oxypurinol | 14.27 (4.119) | 13.41 (2.735)

20. Secondary Outcome: Time of Last Quantifiable Plasma Concentration (Tlast) for Verinurad, M1, M8, Allopurinol, and Oxypurinol
Description: as for outcome 15
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 22 | 24
Hour
  Verinurad | 48.05 [48.00 to 48.13] | 48.07 [48.02 to 48.18]
  M1 | 48.05 [48.00 to 48.13] | 48.07 [48.02 to 48.18]
  M8 | 48.05 [48.00 to 48.13] | 48.07 [48.02 to 48.18]
  Allopurinol | 8.00 [6.00 to 8.02] | 7.03 [6.00 to 8.03]
  Oxypurinol | 48.05 [48.00 to 48.13] | 48.07 [48.02 to 48.18]

21. Secondary Outcome: Apparent Total Body Clearance of Drug From Plasma After Extravascular Administration (Parent Drug Only) (CL/F) for Verinurad and Allopurinol
Description: Assessment of the PK of verinurad and allopurinol in healthy participants.
Time Frame: as for outcome 14
Population: The PK Analysis Set consisted of all participants in the Safety Analysis Set for whom at least 1 reportable PK parameter could be calculated and who had no major protocol deviations thought to impact the analysis of the PK data. Here, number analyzed in each row signifies only the participants with available data that were analyzed for Verinurad/allopurinol.
Measure: Mean (Standard Deviation); unit: Liter/Hour
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 22 | 24
Liter/Hour
  Verinurad: number analyzed (Participants) | 20 | 24
  Verinurad | 64.07 (19.43) | 45.09 (13.13)
  Allopurinol | 71.03 (26.45) | 68.08 (21.28)

22. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration (Parent Drug Only) (Vz/F) for Verinurad and Allopurinol
Description: Assessment of the PK of verinurad and allopurinol in healthy participants.
Time Frame: as for outcome 14
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 22 | 24
Liter
  Verinurad: number analyzed (Participants) | 20 | 24
  Verinurad | 1342 (500.1) | 856.1 (413.5)
  Allopurinol | 103.6 (45.48) | 97.96 (28.94)

23. Secondary Outcome: Apparent Volume of Distribution at Steady State Following Extravascular Administration (Parent Drug Only) (Vss/F) for Verinurad and Allopurinol
Description: Assessment of the PK of verinurad and allopurinol in healthy participants.
Time Frame: as for outcome 14
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 22 | 24
Liter
  Verinurad: number analyzed (Participants) | 20 | 24
  Verinurad | 1060 (336.6) | 448.6 (227.5)
  Allopurinol | 182.9 (79.88) | 165.3 (61.06)

24. Secondary Outcome: Mean Residence Time of the Unchanged Drug in the Systemic Circulation From Zero to Infinity (MRT) for Verinurad and Oxypurinol
Description: Assessment of the PK of verinurad and allopurinol in healthy participants.
Time Frame: as for outcome 14
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 22 | 24
Hour
  Verinurad: number analyzed (Participants) | 20 | 24
  Verinurad | 16.47 (26.78) | 9.320 (34.79)
  Allopurinol | 2.517 (24.44) | 2.383 (18.95)

25. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Examination of the safety and tolerability of verinurad and allopurinol.
Time Frame: From Screening (Day -28 to Day -2) until the Follow-up visit (7 to 10 Days After the Last Dose)
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug (verinurad, allopurinol, and placebo) and for whom any safety post-dose data were available.
Measure: Number; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 22 | 24 | 23
Participants
  Any AE | 8 | 4 | 5
  Any AE with outcome = death | 0 | 0 | 0
  Any Serious adverse events (including events with outcome = death) | 0 | 0 | 0
  Any AE leading to discontinuation of study drug | 0 | 1 | 0
  Any AE leading to withdrawal from study | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From Screening (Day -28 to Day -2) until the Follow-up visit (7 to 10 Days After the Last Dose)
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 8/22 | 4/24 | 5/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=22) | Treatment B (N=24) | Treatment C (N=23)
Headache (Nervous system disorders) | 4 | 3 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Medical device site reaction (General disorders) | 1 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca AB.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT04256629/Prot_SAP_000.pdf